CLINICAL TRIAL: NCT00190684
Title: Long-Term, Open Label Safety Study of Atomoxetine Hydrochloride in Patients, 6 Years and Older With Attention-Deficit/Hyperactivity Disorder
Brief Title: Long-Term, Open Label Atomoxetine Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4331; B4Z-MC-LYAI (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2010-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

ARMS (1):
- Atomoxetine (Experimental): Atomoxetine-naive patients will have an acute titration to a stable dose, atomoxetine experienced patients whose therapy has been interrupted with be rapidly titrated to their previously established stable dose, and atomoxetine patients on a known stable dose may continue treatment at that dose.
  Interventions: Drug: atomoxetine

INTERVENTIONS:
Drug: atomoxetine — 0.5-1.8 mg/kg/day, by mouth (PO), for up to 5 years
  Other Names: LY139603; Strattera

SUMMARY:
To learn about the safety and any side effects of atomoxetine when given to children and adolescents for about 5 years (long-term) and to learn whether atomoxetine can help children and adolescents with attention-deficit/hyperactivity disorder (ADHD) who take the drug for about 5 years (long-term).

Study participants can be atomoxetine naive, atomoxetine experienced whose therapy has been interrupted or, atomoxetine experienced on a known stable dose.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 6 years old but less than 18 years old when enrolled in first atomoxetine study
* Must meet the study criteria for ADHD
* Must be willing to have blood drawn and to complete other test required for this study

Exclusion Criteria:

* allergic to more than 1 kind of medicine or have had multiple bad reactions to any drug
* taking certain medicines that could interact with atomoxetine
* plan to move too far away from a doctor participating in this study in the next 5 years
* current or past history of any of the following: alcohol or drug abuse within the past 3 months, bipolar I or II disorder, high blood pressure, organic brain disease or seizures, psychosis, other disorders or conditions diagnosed by a doctor that might make you unsuitable to participate in this study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1553 (Actual)
Dates: Start 2000-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-619-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (99):
- United States (70):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Centro, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Walnut Creek, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norwich, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainsville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tallahassee, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northbrook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bardstown, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moorestown, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piscataway, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manhasset, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Hyde Park, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stony Brook, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hershey, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rydal, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Providence, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galveston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfax, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herndon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midlothian, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marshfield, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleton, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wallsend, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Brisbane, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Perth, Western Australia
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec, Quebec
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heiligenstadt/Ofr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
- Israel (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ness Ziona
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cagliari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utrecht
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oslo, Norway
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benmore, Sandown
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garsfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Panorama
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg, Sweden
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield, South Yorkshire

REFERENCES:
- [Derived] Michelson D, Read HA, Ruff DD, Witcher J, Zhang S, McCracken J. CYP2D6 and clinical response to atomoxetine in children and adolescents with ADHD. J Am Acad Child Adolesc Psychiatry. 2007 Feb;46(2):242-51. doi: 10.1097/01.chi.0000246056.83791.b6. PMID 17242628
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine: Atomoxetine-naive patients will have an acute titration to a stable dose, atomoxetine experienced patients whose therapy has been interrupted will be rapidly titrated to their previously established stable dose, and atomoxetine patients on a known stable dose may continue treatment at that dose.
Period: Overall Study
Arm/Group | Atomoxetine
Started | 1553
Received at Least 1 Dose of Study Drug | 1551 (1553 patients entered the study; 1551 were enrolled and received study drug.)
Completed | 64 (Number of patients that completed overall study (through Period VI))
Not Completed | 1489
Not completed — Adverse Event | 86
Not completed — Satisfactory response | 80
Not completed — Lack of efficacy | 204
Not completed — Lost to Follow-up | 232
Not completed — Patient moved | 60
Not completed — Patient Decision | 432
Not completed — Clinical relapse | 67
Not completed — Sponsor's decision | 17
Not completed — Physician Decision | 84
Not completed — Protocol Violation | 123
Not completed — Study Period III Completed | 103
Not completed — Study Period V Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1553
Age Continuous [Mean (Standard Deviation); unit: years] | 11.62 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 338
  Male | 1215
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1317
  African Descent | 98
  East/ Southeast Asian | 9
  Western Asian | 1
  Hispanic | 76
  Other | 52
Region of Enrollment [Number; unit: participants]
  United States | 1288
  Israel | 16
  United Kingdom | 24
  Italy | 11
  France | 21
  Canada | 14
  Puerto Rico | 19
  Belgium | 20
  Australia | 22
  South Africa | 19
  Germany | 21
  Netherlands | 15
  Norway | 13
  Sweden | 27
  Spain | 23
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Summary of baseline characteristics is based on 1553 participants, but only 1527 participants have non-missing baseline measurement of height.
  centimeters (cm) | 147.89 (15.72)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Summary of baseline characteristics is based on 1553 participants, but only 1548 participants have non-missing baseline measurement of weight.
  kilograms (kg) | 43.73 (16.03)
Attention Deficit Hyperactive Disorder (ADHD) Subtype [Number; unit: participants] — Summary of baseline characteristics is based on 1553 participants, but only 1547 participants have non-missing baseline measurement of ADHD subtype diagnosis.
  participants
    Inattentive | 413
    Hyperactive/Impulsive | 46
    Combined | 1016
    Not Applicable | 72
    Unknown | 6

OUTCOME MEASURES:

1. Primary Outcome: Categorical Changes in Vital Signs (Blood Pressure [BP], Pulse, Weight, Temperature) During the Study
Description: Vital signs were assesed categorically using the term high for BP, high and low for pulse and temperature, or decreased for weight. For BP, high was an increase to a value above the 95th percentile of the National Institute of Health (NIH) values. For pulse, high was an increase of at least 25 beats per minute to at least 110, and low was a decrease of at least 20 beats per minute to at most 65 beats per minute. For temperature, high was an increase of at least 1 to 37.7 and low was a decrease of at least 1.3 to at most 35.6. Decrease in weight was marked by a reduction of at least 3.5%.
Time Frame: Baseline through 5 years
Population: For each vital sign, the number of participants analyzed was defined as all patients with a baseline and post-baseline measurement, except patients reported as not taking any study drug. Number of subject analyzed for each vital sign is provided.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1528
participants
  Systolic BP High (N=1431) | 228
  Diastolic BP High (N=1458) | 92
  Pulse High (N=1528) | 19
  Pulse Low (N=1528) | 39
  Temperature High (N=1525) | 7
  Temperature Low (N=1525) | 9
  Weight Decrease (N=1526) | 61

2. Primary Outcome: Change From Baseline to 5 Year Endpoint in BP
Time Frame: baseline, 5 years
Population: The number of participants analyzed was defined as all patients with a baseline and post-baseline measurement, except patients reported as not taking any study drug.
Measure: Mean (Standard Deviation); unit: millimeters of Mercury (mmHg)
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1528
millimeters of Mercury (mmHg)
  Systolic BP | 4.7 (11.56)
  Diastolic BP | 1.3 (9.04)
Statistical Analysis 1: Comparison: Atomoxetine; Tested was the null hypothesis that there would be no statistically significant difference between baseline and endpoint; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for systolic BP; Change = endpoint-baseline
Statistical Analysis 2: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon sign-rank test — p-value is for diastolic BP; Change = endpoint-baseline

3. Primary Outcome: Change From Baseline to 5 Year Endpoint in Pulse
Time Frame: baseline, 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1528
beats per minute (bpm) | -1.5 (13.83)
Statistical Analysis 1: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for pulse

4. Primary Outcome: Change From Baseline to 5 Year Endpoint in Body Weight
Time Frame: baseline, 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1526
kilograms (kg) | 11.0 (11.66)
Statistical Analysis 1: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for weight

5. Primary Outcome: Change From Baseline to 5 Year Endpoint in Height
Time Frame: baseline, 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1476
centimeters (cm) | 10.9 (10.41)
Statistical Analysis 1: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for height

6. Primary Outcome: Change From Baseline to 5 Year Endpoint in Weight, Height, and Body Mass Index (BMI) Percentile Stratified by Baseline Quartile
Description: Patients were assessed for changes in weight, height, and BMI. BMI is an estimate of body fat based on body weight divided by height squared.
Time Frame: baseline, 5 years
Population: The number of participants analyzed was defined as all patients with a baseline and 5 year endpoint measurement.
Measure: Mean (Standard Deviation); unit: percentiles
Arm/Group | Atomoxetine
Number analyzed (Participants) | 251
percentiles
  Weight (0 to 25th percentile) (N=46) | 18.93 (9.26)
  Weight (25th to 50th percentile) (N=58) | 14.90 (22.31)
  Weight (50th to 75th percentile) (N=50) | -1.33 (20.21)
  Weight (75th to 100th percentile) (N=97) | -6.68 (15.50)
  Height (0 to 25th percentile) (N=64) | 12.06 (21.00)
  Height (25th tp 50th percentile) (N=61) | 9.53 (21.76)
  Height (50th to 75th percentile) (N=55) | -6.28 (22.55)
  Height (75th to 100th percentile) (N=65) | -10.92 (20.31)
  BMI (0 to 25th percentile) (N=34) | 18.71 (24.76)
  BMI (25th to 50th percentile) (N=53) | 8.52 (28.11)
  BMI (50th to 75th percentile) (N=55) | -3.26 (25.69)
  BMI (75th to 100th percentile) (N=101) | -7.94 (18.41)
Statistical Analysis 1: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, paired t-test — p-value is for weight 0 to 25th percentile
Statistical Analysis 2: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, paired t-test — p-value is for weight 25th to 50th percentile
Statistical Analysis 3: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.644, paired t-test — p-value is for weight 50th to 75th percentile
Statistical Analysis 4: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, paired t-test — p-value is for weight 75th to 100th percentile
Statistical Analysis 5: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, paired t-test — p-value is for height 0 to 25th percentile
Statistical Analysis 6: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.001, paired t-test — p-value is for height 25th to 50th percentile
Statistical Analysis 7: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.044, paired t-test — p-value is for height 50th to 75th percentile
Statistical Analysis 8: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, paired t-test — p-value is for height 75th to 100th percentile
Statistical Analysis 9: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, paired t-test — p-value is for BMI 0 to 25th percentile
Statistical Analysis 10: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.032, paired t-test — p-value is for BMI 25th to 50th percentile
Statistical Analysis 11: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.351, paired t-test — p-value is for BMI 50th to 75th percentile
Statistical Analysis 12: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, paired t-test — p-value is for BMI 75th to 100th percentile

7. Primary Outcome: Change From Baseline to 5 Year Endpoint in Electrocardiogram (ECG)
Description: Patients were assessed for changes in ECG. The RR interval is the time duration between two consecutive R waves of the ECG. The QRS interval is the beginning of Q to the end of the S wave. The QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate. A corrected QT interval (QTc) has been corrected in order to aid interpretation. QTbz is the QT interval using Bazett's correction formula. QTfr is the QT interval using Fridericia's correction formula.QTdat is the QT interval using a data specific correction method for children.
Time Frame: baseline, 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1482
milliseconds (msec)
  RR Interval | 27.2 (138.78)
  QRS Interval | 2.6 (7.19)
  QT Bazett (bz) Correction | -1.7 (17.85)
  QT Data (dat) Correction | -0.2 (15.43)
  QT Fridericia (fr) Correction | 0.5 (15.71)
Statistical Analysis 1: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for RR interval
Statistical Analysis 2: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for QRS Interval
Statistical Analysis 3: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for QT Bazett Correction
Statistical Analysis 4: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.310, Wilcoxon signed-rank test — p-value is for QT Data Correction
Statistical Analysis 5: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.632, Wilcoxon signed-rank test — p-value is for QT Fridericia Correction

8. Primary Outcome: Change From Baseline to 5 Year Endpoint in Heart Rate
Description: Patients were assessed for changes in heart rate using electrocardiogram.
Time Frame: baseline, 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1482
beats per minute (bpm) | -2.5 (14.45)
Statistical Analysis 1: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for HR

9. Primary Outcome: Number of Patients Meeting Committee for Proprietary Medicinal Products (CPMP) Categorical QTc Interval Criteria Part I (Numerical Increase)
Description: QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate. A corrected QT interval (QTc) has been corrected in order to aid interpretation. QTbz is the QT interval using Bazett's correction formula. QTfr is the QT interval using Fridericia's correction formula. QTdat is the QT interval using a data specific correction method for children.
Time Frame: baseline through 5 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1482
participants
  QTc (bz) Increase of at least 30 milliseconds (ms) | 68
  QTc (bz) Increase of at least 60 ms | 2
  QTc (bz) Increase to values >500 ms | 0
  QTc (dat) Increase of at least 30 ms | 50
  QTc (dat) Increase of at least 60 ms | 2
  QTc (dat) Increase to values >500 ms | 0
  QTc (fr) Increase of at least 30 ms | 56
  QTc (fr) Increase of at least 60 ms | 2
  QTc (fr) Increase to values >500 ms | 0

10. Secondary Outcome: Change From Baseline to 5 Year Endpoint in Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) Total Score and Subscale Scores
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of ADHD. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54. Hyperactive/Impulsive and Inattention Subscales consisted of 9 items each, for total subscale score range of 0 to 27. ADHD Index Subscale consisted of 12 items, for total score range of 0 to 36.
Time Frame: baseline, 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1135
units on a scale
  Total Score | 3.5 (9.62)
  Inattentive Subscale Score | 2.6 (6.00)
  Hyperactive Subscale Score | 0.9 (4.73)
Statistical Analysis 1: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for Total Score
Statistical Analysis 2: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for Inattentive Subscale Score
Statistical Analysis 3: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for Hyperactive Subscale Score

11. Secondary Outcome: Change From Baseline to 5 Year Endpoint in Clinical Global Impressions-Attention-Deficit/Hyperactivity Disorder-Severity (CGI-ADHD-S) Score
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: baseline, 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1136
units on a scale | 0.523 (1.149)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for CGI ADHD Severity within group; This test is for a significance of a location shift from zero of the change from baseline within a treatment group

12. Secondary Outcome: Change From Baseline to 5 Year Endpoint in Conners' Parent Rating Scale-Revised: Short Form (CPRS-R:S) Subscale Scores
Description: A 27-item rating scale (0 [not at all/never] to 3 [very much true/very often]) completed by the parent to assess problem behaviors related to ADHD. Subscales: Oppositional, Cognitive Problems, Hyperactivity, and ADHD Index. Subscale total scores range from 0 to 18 for all subscales except ADHD Index which ranges from 0 to 36.
Time Frame: baseline, 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1059
units on a scale
  CPRS ADHD Index Subscale (n=1056) | 2.411 (7.785)
  CPRS Cognitive Subscale (n=1056) | 1.500 (4.777)
  CPRS Hyperactive Subscale (n=1057) | 0.325 (3.287)
  CPRS Oppositional Subscale (n=1059) | 1.357 (4.287)
Statistical Analysis 1: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for CPRS ADHD Index Subscale within group; This test is for a significance of a location shift from zero of the change from baseline within a treatment group
Statistical Analysis 2: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for CPRS Cognitive Subscale; This test is for a significance of a location shift from zero of the change from baseline within a treatment group
Statistical Analysis 3: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.026, Wilcoxon signed-rank test — p-value is for CPRS Hyperactive Subscale; This test is for a significance of a location shift from zero of the change from baseline within a treatment group
Statistical Analysis 4: Comparison: Atomoxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — p-value is for CPRS Oppositional Subscale; This test is for a significance of a location shift from zero of the change from baseline within a treatment group

13. Secondary Outcome: Change From Baseline to 5 Year Endpoint in the Stroop Word Color Test
Description: Only patients who took the Stroop Color Word Test in a previous atomoxetine study were required to complete the Stroop in this study. Stroop measures inhibition of dominant response and interference control. Patients were given tasks of recognition (colors), reading (where a word represents a color), and interference (reading words written in different colors). There were 100 items for each of the three categories and if they made it through 100 words with time remaining, they would repeat the list. Only a small number of patients had Stroop tests in this study, so no analysis was done.
Time Frame: baseline, 5 years
Population: There were not enough participants with prior Stroop Word Color tests to analyze the data.
Measure: Mean (Standard Deviation); unit: number of correct answers
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

14. Primary Outcome: Number of Patients Meeting CPMP Categorical QTc Interval Criteria Part II (Interpretation at Baseline and Endpoint)
Description: QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate. A corrected QT interval (QTc) has been corrected in order to aid interpretation. QTbz is the QT interval using Bazett's correction formula. QTfr is the QT interval using Fridericia's correction formula. QTdat is the QT interval using a data specific correction method for children. For Males: Normal is <430 ms, Borderline is >=430 ms and <450 ms, Prolonged is >=450 ms. For Females: Normal is <450 ms, Borderline is >=450 ms and <470 ms, Prolonged is >=470 ms.
Time Frame: baseline through 5 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1482
participants
  QTc (bz) Normal Baseline/Normal Endpoint | 1069
  QTc (bz) Normal Baseline/Borderline Endpoint | 156
  QTc (bz) Normal Baseline/Prolonged Endpoint | 11
  QTc (bz) Borderline Baseline/Normal Endpoint | 180
  QTc (bz) Borderline Baseline/Borderline Endpoint | 49
  QTc (bz) Borderline Baseline/Prolonged Endpoint | 6
  QTc (bz) Prolonged Baseline/Normal Endpoint | 6
  QTc (bz) Prolonged Baseline/Borderline Endpoint | 5
  QTc (bz) Prolonged Baseline/Prolonged Endpoint | 0
  QTc (dat) Normal Baseline/Normal Endpoint | 1433
  QTc (dat) Normal Baseline/Borderline Endpoint | 26
  QTc (dat) Normal Baseline/Prolonged Endpoint | 1
  QTc (dat) Borderline Baseline/Normal Endpoint | 16
  QTc (dat) Borderline Baseline/Borderline Endpoint | 3
  QTc (dat) Borderline Baseline/Prolonged Endpoint | 1
  QTc (dat) Prolonged Baseline/Normal Endpoint | 2
  QTc (dat) Prolonged Baseline/Borderline Endpoint | 0
  QTc (dat) Prolonged Baseline/Prolonged Endpoint | 0
  QTc (fr) Normal Baseline/Normal Endpoint | 1454
  QTc (fr) Normal Baseline/Borderline Endpoint | 16
  QTc (fr) Normal Baseline/Prolonged Endpoint | 2
  QTc (fr) Borderline Baseline/Normal Endpoint | 7
  QTc (fr) Borderline Baseline/Borderline Endpoint | 0
  QTc (fr) Borderline Baseline/Prolonged Endpoint | 1
  QTc (fr) Prolonged Baseline/Normal Endpoint | 2
  QTc (fr) Prolonged Baseline/Borderline Endpoint | 0
  QTc (fr) Prolonged Baseline/Prolonged Endpoint | 0

15. Primary Outcome: Number of Participants With Abnormal Laboratory Analytes During the Study
Description: Standard reference ranges from Covance Laboratories were used in the determination of abnormal high and low values based on age and gender, where appropriate. Aspartate aminotransferase (AST); serum glutamic oxaloacetic transaminase (SGOT); units/liter (U/L); alanine aminotransferase (ALT); serum glutamic pyruvic transaminase (SGPT); millimoles/liter (mmol/L); grams/liter (g/L); micromoles/liter (umol/L); millimoles/liter-iron (mmol/L-Fe); trillion/liter (TI/L)or 10^12 units/liter; Giga/liter (GI/L)or 10^9 units/liter; femtoliters (fL); urinalysis (UA)
Time Frame: baseline through 5 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 1487
participants
  AST/SGOT (U/L) Low (N=1484) | 0
  AST/SGOT (U/L) High (N=1484) | 27
  ALT/SGPT (U/L) Low (N=1486) | 2
  ALT/SGPT (U/L) High (N=1486) | 38
  Creatine Phosphokinase (U/L) Low (N=1485) | 0
  Creatine Phosphokinase (U/L) High (N=1485) | 57
  Alkaline Phosphatase (U/L) Low (N=1486) | 67
  Alkaline Phosphatase (U/L) High (N=1486) | 83
  Gamma Glutamyltransferase (U/L) Low (N=1486) | 0
  Gamma Glutamyltransferase (U/L) High (N=1486) | 17
  Urea Nitrogen (mmol/L) Low (N=1487) | 1
  Urea Nitrogen (mmol/L) High (N=1487) | 2
  Calcium (mmol/L) Low (N=1487) | 0
  Calcium (mmol/L) High (N=1487) | 117
  Inorganic Phosphorus (mmol/L) Low (N=1485) | 10
  Inorganic Phosphorus (mmol/L) High (N=1485) | 31
  Total Protein (g/L) Low (N=1487) | 2
  Total Protein (g/L) High (N=1487) | 5
  Albumin (g/L) Low (N=1487) | 1
  Albumin (g/L) High (N=1487) | 113
  Glucose, Non-Fasting/Random (mmol/L) Low (N=1486) | 20
  Glucose, Non-Fasting/Random (mmol/L) High (N=1486) | 1
  Uric Acid (umol/L) Low (N=1487) | 6
  Uric Acid (umol/L) High (N=1487) | 130
  Cholesterol (mmol/L) Low (N=1487) | 87
  Cholesterol (mmol/L) High (N=1487) | 72
  Creatinine (umol/L) Low (N=1487) | 0
  Creatinine (umol/L) High (N=1487) | 285
  Total Bilirubin (umol/L) Low (N=1458) | 0
  Total Bilirubin (umol/L) High (N=1458) | 38
  Hematocrit (1) Low (N=1482) | 24
  Hematocrit (1) High (N=1482) | 85
  Hemoglobin (mmL/L-Fe) Low (N=1482) | 14
  Hemoglobin (mmL/L-Fe) High (N=1482) | 30
  Erythrocyte Count (TI/L) Low (N=1482) | 8
  Erythrocyte Count (TI/L) High (N=1482) | 3
  Leukocyte Count (GI/L) Low (N=1482) | 63
  Leukocyte Count (GI/L) High (N=1482) | 8
  Bands (GI/L) Low (N=1482) | 0
  Bands (GI/L) High (N=1482) | 0
  Neutrophils, Segmented (GI/L) Low (N=1482) | 20
  Neutrophils, Segmented (GI/L) High (N=1482) | 23
  Lymphocytes (GI/L) Low (N=1482) | 6
  Lymphocytes (GI/L) High (N=1482) | 0
  Monocytes (GI/L) Low (N=1482) | 62
  Monocytes (GI/L) High (N=1482) | 12
  Eosinophils (GI/L) Low (N=1482) | 0
  Eosinophils (GI/L) High (N=1482) | 54
  Basophils (GI/L) Low (N=1482) | 0
  Basophils (GI/L) High (N=1482) | 3
  Mean Cell Volume (fL) Low (N=1482) | 26
  Mean Cell Volume (fL) High (N=1482) | 10
  Platelet Count (GI/L) Low (N=1479) | 1
  Platelet Count (GI/L) High (N=1479) | 63
  Sodium (mmol/L) Low (N=1486) | 0
  Sodium (mmol/L) High (N=1486) | 2
  Potassium (mmol/L) Low (N=1484) | 0
  Potassium (mmol/L) High (N=1484) | 8
  Chloride (mmol/L) Low (N=1486) | 0
  Chloride (mmol/L) High (N=1486) | 2
  Bicarbonate (mmol/L) Low (N=1486) | 7
  Bicarbonate (mmol/L) High (N=1486) | 6
  UA-Specific Gravity (no units) Low (N=1486) | 39
  UA-Specific Gravity (no units) High (N=1486) | 73
  Lymphocytes, Atypical (GI/L) Low (N=52) | 0
  Lymphocytes, Atypical (GI/L) High (N=52) | 52

16. Primary Outcome: Number of Participants in Each Tanner Stage (Pubic Hair) by Age Group
Description: Tanner Stage:
  I: no pubic hair at all (prepubertal Dominic state) II: small amount of long, downy hair with slight pigmentation at the base of the penis and scrotum (males) or on the labia majora (females) III: hair becomes more coarse and curly, and begins to extend laterally IV: adult-like hair quality, extending across pubis but sparing medial thighs V: hair extends to medial surface of the thighs
  Age Groups:
  1. age<11.0 (female) and age<12 (male)
  2. 11=<age<12 (female) or 12<=age<13 (male)
  3. 12=<age<15 (female) or 13=<age<15 (male)
  4. age>=15 (female and male)
Time Frame: 1 year through 5 years
Population: The analysis population is defined as patients with at least two Tanner measurements.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 93
participants
  First Tanner, Age Group 1, Tanner I (N=7) | 2
  First Tanner, Age Group 1, Tanner II (N=7) | 2
  First Tanner, Age Group 1, Tanner III (N=7) | 2
  First Tanner, Age Group 1, Tanner IV (N=7) | 1
  First Tanner, Age Group 1, Tanner V (N=7) | 0
  First Tanner, Age Group 2, Tanner I (N=14) | 4
  First Tanner, Age Group 2, Tanner II (N=14) | 6
  First Tanner, Age Group 2, Tanner III (N=14) | 2
  First Tanner, Age Group 2, Tanner IV (N=14) | 2
  First Tanner, Age Group 2, Tanner V (N=14) | 0
  First Tanner, Age Group 3, Tanner I (N=37) | 0
  First Tanner, Age Group 3, Tanner II (N=37) | 2
  First Tanner, Age Group 3, Tanner III (N=37) | 13
  First Tanner, Age Group 3, Tanner IV (N=37) | 15
  First Tanner, Age Group 3, Tanner V (N=37) | 7
  First Tanner, Age Group 4, Tanner I (N=35) | 0
  First Tanner, Age Group 4, Tanner II (N=35) | 0
  First Tanner, Age Group 4, Tanner III (N=35) | 2
  First Tanner, Age Group 4, Tanner IV (N=35) | 11
  First Tanner, Age Group 4, Tanner V (N=35) | 22
  Endpoint Tanner, Age Group 1, Tanner I (N=2) | 1
  Endpoint Tanner, Age Group 1, Tanner II (N=2) | 1
  Endpoint Tanner, Age Group 1, Tanner III (N=2) | 0
  Endpoint Tanner, Age Group 1, Tanner IV (N=2) | 0
  Endpoint Tanner, Age Group 1, Tanner V (N=2) | 0
  Endpoint Tanner, Age Group 2, Tanner I (N=4) | 0
  Endpoint Tanner, Age Group 2, Tanner II (N=4) | 1
  Endpoint Tanner, Age Group 2, Tanner III (N=4) | 2
  Endpoint Tanner, Age Group 2, Tanner IV (N=4) | 1
  Endpoint Tanner, Age Group 2, Tanner V (N=4) | 0
  Endpoint Tanner, Age Group 3, Tanner I (N=32) | 0
  Endpoint Tanner, Age Group 3, Tanner II (N=32) | 5
  Endpoint Tanner, Age Group 3, Tanner III (N=32) | 8
  Endpoint Tanner, Age Group 3, Tanner IV (N=32) | 14
  Endpoint Tanner, Age Group 3, Tanner V (N=32) | 5
  Endpoint Tanner, Age Group 4, Tanner I (N=55) | 0
  Endpoint Tanner, Age Group 4, Tanner II (N=55) | 0
  Endpoint Tanner, Age Group 4, Tanner III (N=55) | 3
  Endpoint Tanner, Age Group 4, Tanner IV (N=55) | 19
  Endpoint Tanner, Age Group 4, Tanner V (N=55) | 33

ADVERSE EVENTS:
Arm/Group | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 92/1551
Other Adverse Events (participants affected / at risk) | 1372/1551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=1551)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 10 (10)
Campylobacter infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (4)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Sinusitis (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 2 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 4 (4)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (5)
Blood pressure decreased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (10)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Retrognathia (Musculoskeletal and connective tissue disorders) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Complex partial seizures (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Migraine with aura (Nervous system disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 3 (5)
Agitation (Psychiatric disorders) | 1 (1)
Conduct disorder (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 5 (5)
Impulsive behaviour (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Negativism (Psychiatric disorders) | 1 (1)
Oppositional defiant disorder (Psychiatric disorders) | 1 (2)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Pyromania (Psychiatric disorders) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 9 (9)
Suicide attempt (Psychiatric disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Facial operation (Surgical and medical procedures) | 1 (1)
Nasal septal operation (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=1551)
Abdominal pain (Gastrointestinal disorders) | 82 (100)
Abdominal pain upper (Gastrointestinal disorders) | 260 (353)
Diarrhoea (Gastrointestinal disorders) | 125 (166)
Nausea (Gastrointestinal disorders) | 210 (285)
Vomiting (Gastrointestinal disorders) | 285 (451)
Fatigue (General disorders) | 147 (186)
Irritability (General disorders) | 151 (168)
Pyrexia (General disorders) | 248 (386)
Seasonal allergy (Immune system disorders) | 89 (98)
Ear infection (Infections and infestations) | 79 (108)
Gastroenteritis viral (Infections and infestations) | 122 (152)
Influenza (Infections and infestations) | 205 (287)
Nasopharyngitis (Infections and infestations) | 315 (515)
Pharyngitis streptococcal (Infections and infestations) | 129 (177)
Sinusitis (Infections and infestations) | 125 (176)
Upper respiratory tract infection (Infections and infestations) | 263 (430)
Viral infection (Infections and infestations) | 78 (106)
Decreased appetite (Metabolism and nutrition disorders) | 163 (178)
Dizziness (Nervous system disorders) | 83 (103)
Headache (Nervous system disorders) | 534 (1063)
Depression (Psychiatric disorders) | 81 (84)
Insomnia (Psychiatric disorders) | 106 (120)
Cough (Respiratory, thoracic and mediastinal disorders) | 297 (445)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 79 (97)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 168 (263)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 267 (414)
Acne (Skin and subcutaneous tissue disorders) | 105 (110)
Rash (Skin and subcutaneous tissue disorders) | 80 (90)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days